CLINICAL TRIAL: NCT07051330
Title: The Advancing Dynamic And Personalized Training Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: Templeton World Charity Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Other
Other Study IDs: 2025-0660; A171600 (Other: UW Madison)
Record Dates: First submitted 2025-06-24; First posted 2025-07-04 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-09

CONDITIONS: Well-Being, Psychological
Keywords: personalized well-being; HMP app; Healthy Minds Program
MeSH Terms: conditions — Psychological Well-Being | interventions — Amyloid

STUDY DESIGN:
Intervention Model Description: Participants are randomized to six different binary conditions. The investigators plan to collapse the groups for analysis, for example, combining participants with or without the introduction videos, regardless of their other assigned conditions.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Introduction Video to HMP app (Experimental): All participants are randomized to this condition (Yes or No)
  Interventions: Other: Healthy Minds Program (HMP) app
- Introduction Video to Training Modules (Experimental): All participants are randomized to this condition (Yes or No)
  Interventions: Other: Healthy Minds Program (HMP) app
- Module Order based on ACIP Score (Experimental): All participants are randomized to this condition (Highest score first or Lowest score first)
  Interventions: Other: Healthy Minds Program (HMP) app
- Practice-Nudging Test Messages (Experimental): All participants are randomized to this condition (Yes or No)
  Interventions: Other: Healthy Minds Program (HMP) app
- Microsupport Messages During Intervention (Experimental): All participants are randomized to this condition (Yes or No)
  Interventions: Other: Healthy Minds Program (HMP) app
- Microsupport Messages During Follow-Up (Experimental): All participants are randomized to this condition (Yes or No)
  Interventions: Other: Healthy Minds Program (HMP) app

INTERVENTIONS:
Other: Healthy Minds Program (HMP) app — All participants will complete baseline surveys, weekly questionnaires (for 4 weeks) through the HMP app intervention, and will be surveyed again at 3-months post-intervention. Participants are randomized to each of the following binary conditions.
  1. Introduction video for the app (yes / no)
  2. Introduction video for the training modules (yes / no)
  3. Module order based on ACIP score (highest-first / lowest-first)
  4. Practice-nudging text messages (yes / no)
  5. Microsupport messages during the intervention period (yes / no)
  6. Microsupport messages during the follow-up period (yes / no
  Other Names: HMP app

SUMMARY:
This study aims to enhance the Healthy Minds Program (HMP) app by developing and testing a personalized, data-driven approach to optimize long-term well-being. 1100 participants will be enrolled and on study for up to 4 months (4 week intervention plus 3 month follow-up).

DETAILED DESCRIPTION:
Participants will be randomly assigned to various training conditions that vary across six factors. Each of the six factors is binary ("yes" vs. "no"), and for each factor there is a 50 percent probability of assignment to either level.

1. Introduction video for the app (yes / no)
2. Introduction video for the training modules (yes / no)
3. Module order based on ACIP score (highest-first / lowest-first)
4. Practice-nudging text messages (yes / no)
5. Microsupport messages during the intervention period (yes / no)
6. Microsupport messages during the follow-up period (yes / no)

Participants will take surveys at baseline, weekly through the 4-week intervention, and 3-month follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Elevated symptoms of depression (PHQ-9 greater than or equal to 5)
* proficiency in English
* access to a smartphone and internet
* ability to receive text messages

Exclusion Criteria:

* Prior experience with meditation
* Prior use of the Healthy Minds Program app
* History of psychosis or mania
* Plans to travel in the next six weeks
* Suicidal ideation or thoughts of self-harm indicated by PHQ-9 item 9 and BDI item 9
* Failure to select the correct code word mentioned in the welcome video
* Not a US citizen
* Non-permanent resident
* Self-identification as artificial intelligence (AI)
* Has a hearing impairment

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1500 (Estimated)
Dates: Start 2025-07-20 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Change in PHQ-9 | Baseline, week 1, week 2, week 3, week 4 (of intervention period), and 3 month follow-up (up to 4 months on study)
  PHQ-9 is a 9 item questionnaire where participants report how often in the past 2 weeks they were bothered by specific problems. It is scored on a 4-point Likert scale, where 0=not at all and 4=nearly every day. Scores range from 0-36, where higher scores indicate more depressive symptoms.

SECONDARY OUTCOMES:
Change in Patient-Reported Outcomes Measurement Information System (PROMIS) Depression | Baseline, week 1, week 2, week 3, week 4 (of intervention period), and 3 month follow-up (up to 4 months on study)
  A computer-adaptive measure of feelings of depression scored from 1 to 5 where higher numbers indicate increased feelings of depression. It provides t-scores with a mean of 50 and SD of 10.
Change in PROMIS Anxiety Score | Baseline, week 1, week 2, week 3, week 4 (of intervention period), and 3 month follow-up (up to 4 months on study)
  The PROMIS Anxiety Score is a computer adaptive measure of feelings of anxiety in the past 7 days. This is a computer-adaptive survey scored on a 5-point Likert scale from 1 (never) to 5 (always) with higher scores indicating increased anxiety. It provides t-scores with a mean of 50 and SD of 10. Higher t-scores indicate higher levels of anxiety.
Acceptability of Intervention Measure | week 4 (of intervention period)
  The Acceptability of Intervention Measure is a 4-item self-report measure scored on a 5-point Likert scale. Scores range from 1 (completely disagree) to 5 (completely agree), with higher scores indicating more acceptability of the intervention.
Change in Growth Mindset Scale for Well-Being | Baseline, week 4 (of intervention period), and 3 month follow-up (up to 4 months on study)
  A measure of fixed versus incremental mindset regarding well-being. The average across items for a possible range in scores from 1-6 will be measured, with higher scores indicating greater levels of incremental views on well-being (i.e., it can be learned).
HMP engagement measure | Week 4 (of intervention period), and 3 month follow-up (up to 4 months on study)
  HMP engagement is a 16-item measure which assess participant's usage experience with the Healthy Minds Program. It is scored on a 5-point Likert scale where 1 = Strongly disagree to 5 = Strongly agree. The total possible range of scores is 0-80 where higher scores indicate more positive engagement with the app.
Change in Cannabis Use Disorder Identification Test - Revised (CUDIT-R) | Baseline, week 4 (of intervention period), and 3 month follow-up (up to 4 months on study)
  CUDIT-R is an 8-item survey asking about the participant's relationship to cannabis. It is scored using various scales depending on the item. Scores range from 0 to 32, with higher scores indicating greater risk for cannabis use disorder.
Change in Alcohol Use Disorders Identification Test (AUDIT) | Baseline, week 4 (of intervention period), and 3 month follow-up (up to 4 months on study)
  AUDIT is a 10-item survey asking about the participant's relationship to alcohol. It is scored using various scales depending on the item. Scores range from 0 to 40, with higher scores indicating greater risk for alcohol use disorder.
Change in Healthy Minds Index (HMI) Score | Baseline, week 4 (of intervention period), and 3 month follow-up (up to 4 months on study)
  HMI is a 17-item survey scored on a 5-point Likert scale from 0 (never, none, not at all) to 4 (always, every time, to the highest degree) that assesses awareness, connection, insight, and purpose. Higher scores indicate higher sense of awareness, connection, insight, and purpose. Mean score for each subscale will be reported.
Change in PROMIS Global Health Score | Baseline, week 4 (of intervention period), and 3 month follow-up (up to 4 months on study)
  Global Health is a participant-reported outcome measure that assesses an individual's overall physical and mental health, including their perceptions of general health. It comprises 10 items, with four items assessing Global Physical Health and four assessing Global Mental Health, all based on five core PROMIS domains: physical function, pain, fatigue, emotional distress, and social health. The scores, ranging from 0 to 20, represent the individual's perception of their health, with lower scores indicating greater impairment.
Change in Ruminative Response Scale (RSS) Score | Baseline, week 4 (of intervention period), and 3 month follow-up (up to 4 months on study)
  The RRS is a 10-item, 4-point measure of rumination. Each item indicates the frequency of each event by rating a four-point Likert scale ranging from 1 (Almost never) to 4 (Almost always). The total score ranges from 10-40, with higher scores indicating increased tendency to ruminate.
Change in Big Five Inventory-2 Extra Short Form (BFI-2-XS) | Baseline, week 4 (of intervention period), and 3 month follow-up (up to 4 months on study)
  BFI-2-XS is a 15-item questionnaire designed to assess the Big Five personality domains: Extraversion; Agreeableness; Conscientiousness; Negative Emotionality; and, Open-Mindedness. Each trait is assessed with three items, and the total score for each trait ranges from 3 to 15, with higher scores indicating a stronger tendency towards that trait.
Change in Mindfulness Adherence Questionnaire (MAQ) | Week 4 (of intervention period), and 3 month follow-up (up to 4 months on study)
  MAQ is a 12-item self-report scale designed to assess both the quantity and quality of mindfulness-based practice (MBP), including formal and informal practices. Two items assess the duration of formal practice. The remaining ten items use a 7-point Likert scale ranging from 0 (Never) to 6 (Always) to measure these aspects of mindfulness practice. Scores range from 0-60. Higher scores on the MAQ generally indicate higher levels of practice and/or better quality of practice.
Change in Self-Compassion Scale - Short Form (SCS-SF) | Baseline, week 1, week 2, week 3, week 4 (of intervention period), and 3 month follow-up (up to 4 months on study)
  SCS-SF is a 12-item survey asking how the participant relates to themself. It is scored on a 5-point Likert scale, where 1 = Almost never and 5 = Almost always. Scores range from 12-60, with higher scores indicating greater self-compassion.
Change in Flourishing Index Score | Baseline, week 1, week 2, week 3, week 4 (of intervention period), and 3 month follow-up (up to 4 months on study)
  The Flourishing Index is a 10-item questionnaire where participants report their general level of flourishing (e.g., well-being, health, etc.). It is scored on a 0 to 10-point scale, with anchors varying across items. The total score ranges from 0 to 100 with higher scores indicating higher flourishing.
Change in Digital Working Alliance Inventory (DWAI) | week 1, week 2, week 3, week 4 (of intervention period), and 3 month follow-up (up to 4 months on study)
  DWAI is a six-item questionnaire designed to assess the therapeutic alliance within the Healthy Minds Program (HMP) app. It measures the user's connection and agreement with the app, focusing on the bond, tasks, and goals of the therapeutic relationship. It is scored on a 7-point Likert scale, with scores ranging from 6-42. Higher scores indicate a stronger working alliance with the HMP app.
Change PROMIS Sleep Disturbance Score | Baseline, week 1, week 2, week 3, week 4 (of intervention period), and 3 month follow-up (up to 4 months on study)
  The PROMIS Sleep Disturbance Score is a measure of sleep in the past 7 days. This is a computer-adaptive survey scored on a 5-point Likert scale with higher scores indicating increased sleep disturbance. It provides t-scores with a mean of 50 and SD of 10. Higher t scores indicate higher levels of sleep disturbances.
Change in PROMIS Meaning and Purpose Score | Baseline, week 1, week 2, week 3, week 4 (of intervention period), and 3 month follow-up (up to 4 months on study)
  The PROMIS Meaning and Purpose is a computer-adaptive measures which assesses one's sense of life having purpose and that there are good reasons for living. It is scored on a 5-point Likert scale where 1 = strongly disagree to 5 = strongly agree. Higher scores indicate hopefulness, optimism, goal-directedness, and feelings that one's life is worthy. It provides t-scores with a mean of 50 and a standard deviation of 10 in the general population.
Change in Decentering Subscale of Experiencing Questionnaire score | Baseline, week 1, week 2, week 3, week 4 (of intervention period), and 3 month follow-up (up to 4 months on study)
  The Decentering subscale of the Experience Questionnaire is an 11-item questionnaire where participants report on their ability to decenter from their experience. It is scored on a 5-point Likert scale where 1 = never to 5 = all the time. The total possible range of scores is 11-55 where higher scores indicate a greater ability to decenter from experience.
Change in NIH Toolbox Loneliness Score | Baseline, week 1, week 2, week 3, week 4 (of intervention period), and 3 month follow-up (up to 4 months on study)
  The NIH Toolbox Loneliness is a 5-item questionnaire where participants report how often in the past week they have felt loneliness. It is scored on a 5-point Likert scale where 1 = never to 5 = always. The total possible range of scores is 5-25 where higher scores indicate a greater sense of loneliness.
Change in Five-facet Mindfulness Questionnaire: Awareness Subscale (FFMQ-Acting with Awareness) Score | Baseline, week 1, week 2, week 3, week 4 (of intervention period), and 3 month follow-up (up to 4 months on study)
  The FFMQ-Acting with Awareness subscale is an 8-item survey scored on a 5-point Likert scale from 'never, or very rarely true' to 'very often or always true', for a total possible range of scores from 8-40 where higher scores indicate greater mindfulness awareness.
Change in Five-facet Mindfulness Questionnaire: Non-reactivity Subscale (FFMQ-Non-reactivity) Score | Baseline, week 1, week 2, week 3, week 4 (of intervention period), and 3 month follow-up (up to 4 months on study)
  The FFMQ- Non-reactivity subscale is a 7-item survey scored on a 5-point Likert scale from 1 = 'never, or very rarely true' to 5 = 'very often or always true', for a total possible range of scores from 7-35 where higher scores indicate greater ability to actively detach from negative thoughts and emotions.
Change in Perceived Stress Scale (PSS) Score | Baseline, week 1, week 2, week 3, week 4 (of intervention period), and 3 month follow-up (up to 4 months on study)
  PSS is a 10-item survey scored on a 5-point Likert scale from 0 = never to 4 = very often, for a total possible range of scores from 0-40 where higher scores indicate higher perceived stress.
Morning Daily Diary Items | Daily through the Intervention Period (up to 4 weeks)
  Morning daily diary will include single-item measures of mindfulness, decentering, connection, purpose, depression, anxiety, happiness, energy, stress, busyness, rumination (2 items), sleep quality, motivation to practice meditation, and expectations and challenges related to using the HMP. Each item will be rated on a 5-point Likert scale (1 = not at all, 5 = very much). Higher scores indicate greater levels of the respective construct, such as higher mindfulness, greater decentering, stronger sense of purpose, greater happiness, more severe depression or anxiety, better sleep quality, or greater motivation and perceived helpfulness or frustration with HMP use that morning.
Evening Daily Diary Items | Daily through the Intervention Period (up to 4 weeks)
  Evening daily diary will include single-item measures of mindfulness, decentering, connection, purpose, depression, anxiety, happiness, energy, happy event, stress exposure, rumination (2 items), and expectations related to using the HMP. Each item will be rated on a 5-point Likert scale (1 = not at all, 5 = very much). Higher scores indicate greater levels of the respective construct, such as higher mindfulness, greater decentering, stronger sense of purpose, more severe depression or anxiety, happy event and stressor exposure experience, or greater motivation and perceived helpfulness with HMP use that day.
Percentage of participants with a formal practice | Daily through the Intervention Period (up to 4 weeks)
  Participants' engagement in formal mindfulness practice will be assessed twice a day with a binary yes/no response.
Percentage of participants with a informal practice | Daily through the Intervention Period (up to 4 weeks)
  Participants' engagement in informal mindfulness practice will be assessed twice a day with a 5-point Likert scale (1 = not at all, 5 = all day long).
Percentage of participants received a text message | Daily through the Intervention Period (up to 4 weeks)
  Participants will indicate whether they received a text message from the study that day (yes/no). If they respond "yes," they will then report whether the message encouraged them to apply a wellbeing strategy (yes/no) and rate the extent to which they applied the strategy in their day-to-day activities on a 5-point Likert scale (1 = not at all, 5 = very much).

OTHER OUTCOMES:
Change in Beck Depression Inventory Item 9 Score | Baseline, week 1, week 2, week 3, week 4 (of intervention period), and 3 month follow-up (up to 4 months on study)
  Item 9 on the Beck Depression Inventory (BDI) assesses suicidal thoughts or wishes. The possible scores for this item are 0, 1, 2, or 3, corresponding to different levels of severity. A score of 0 indicates no suicidal thoughts, while higher scores indicate increasing severity of suicidal ideation.
Change in Mindfulness-Based Program - Meditation-Related Adverse Effects Scale (MBP-MRAES) | week 4 (of intervention period), and 3 month follow-up (up to 4 months on study)
  MBP-MRAES is an 11-item questionnaire which measures distressing experiences associated with meditation practice. The first ten items use a frequency-based scale with the following response options: Never, A few days to 1 week, 1 week to 1 month, 1 month to 1 year, and 1 year or longer. If a participant selects any response other than Never, they are prompted with a follow-up question asking them to rate the experience on a scale from Very distressing to Very positive. The eleventh item is an open-ended question that invites participants to describe any other significant symptoms they may have experienced.
Lasting Effects Questionnaire | 3-month follow-up (up to 4 months on study)
  An item about lasting bad effects from the HMP app will be scored on a 5-point scale from 1 = strongly disagree to 5 = strongly agree.
Medication and Therapy Questionnaire | Baseline, week 4 (of intervention period), and 3-month follow-up (up to 4 months on study)
  The 3-item Medication and Therapy Questionnaire collects information on whether participants received medication or therapy for mental health concerns in the past month. Each item is a yes/no question.
Change in Meditation and App Usage | Baseline, week 4 (of intervention period), and 3-month follow-up (up to 4 months on study)
  The 5-item Meditation and App usage Questionnaire assesses participants' engagement with meditation-related activities over two timeframes: the past month (at Week 4) and the past three months (at the 3-month follow-up). Three items ask whether participants used a meditation app, meditated with others, or attended a meditation class or group. Two additional items gather details about the specific meditation app used and the frequency of its use.
Hospitalization | Week 1, week 2, week 3, week 4 (of intervention period), and 3 month follow-up (up to 4 months on study)
  The hospitalization form collects participants' hospitalization history since last survey.

CONTACTS AND LOCATIONS:
Overall Officials: Simon Goldberg, PhD, Principal Investigator — Center for Healthy Minds
Locations (1):
- Center for Healthy Minds, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified data will be shared electronically (e.g., posted on the Open Science Framework). Confidentiality will be protected by stripping the data of all identifiers, including HIPAA identifiers.